CLINICAL TRIAL: NCT01069354
Title: Evaluation of Pain With the Use of Radiesse® With Lidocaine for the Treatment of Nasolabial Folds
Brief Title: Evaluation of Pain With Radiesse® With Lidocaine for Nasolabial Folds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P120677
Record Dates: First submitted 2010-02-15; First posted 2010-02-17 (Estimated); Results first posted 2018-05-30 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2017-09

CONDITIONS: Nasolabial Folds
Keywords: Moderate to severe wrinkles and folds such as nasolabial folds

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radiesse® Mixed with Lidocaine (Experimental): Injectable Dermal Filler. The same participants received the experimental device and the active comparator device at the same time (left and right sides of face).
  Interventions: Device: Radiesse® Injectable Dermal Filler with Lidocaine
- Radiesse® without Lidocaine (Active Comparator): Injectable Dermal Filler. The same participants received the experimental device and the active comparator device at the same time (left and right sides of face).
  Interventions: Device: Radiesse® Injectable Dermal Filler without Lidocaine

INTERVENTIONS:
Device: Radiesse® Injectable Dermal Filler with Lidocaine — Calcium hydroxylapatite particles suspended in an aqueous-based gel carrier with 3% lidocaine hydrochloride (HCl)
  Arms: Radiesse® Mixed with Lidocaine
Device: Radiesse® Injectable Dermal Filler without Lidocaine — Calcium hydroxylapatite particles suspended in an aqueous-based gel carrier without 3% lidocaine hydrochloride (HCl)
  Arms: Radiesse® without Lidocaine

SUMMARY:
To assess pain during nasolabial fold treatment using Radiesse® Injectable Dermal Filler with lidocaine

DETAILED DESCRIPTION:
To assess pain immediately after nasolabial fold treatment with Radiesse® Injectable Dermal Filler with lidocaine in one nasolabial fold compared to Radiesse® Injectable Dermal Filler without lidocaine in the contralateral nasolabial fold

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years of age
* Is a candidate for nasolabial fold treatment using Radiesse
* Has approximately symmetrical nasolabial folds
* Understands and accepts the obligation not to receive any other facial procedures in the lower half of the face for 1 month

Exclusion Criteria:

* Has received any type of treatment or procedures including surgery in the nasolabial folds
* Has received neurotoxin, hyaluronic acid, calcium hydroxylapatite (CaHA) or collagen injections in the lower half of the face within past 6 months
* Has received polylactic acid, polymethyl methacrylate (PMMA), silicone or any other permanent filler in the lower half of the face
* Has nasolabial folds that are too severe to be corrected in one treatment session
* Has any history of hypersensitivity to lidocaine or anesthetics of the amide type

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2012-11; Primary Completion 2013-05 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fred Derosier, DO, Study Director — Merz North America, Inc.
Locations (2):
- Canada (2):
  - Toronto
  - Woodbridge

REFERENCES:
- [Result] Schachter D, Bertucci V, Solish N. Calcium Hydroxylapatite With Integral Lidocaine Provides Improved Pain Control for the Correction of Nasolabial Folds. J Drugs Dermatol. 2016 Aug 1;15(8):1005-10. PMID 27538003

RESULTS

PARTICIPANT FLOW:
Groups:
- Radiesse® Mixed With Lidocaine and Radiesse® Without Lidocaine: Injectable Dermal Filler. The same 102 participants received the experimental device and the active comparator device at the same time (left and right sides of face).
  Calcium hydroxylapatite particles suspended in an aqueous-based gel carrier containing 3% lidocaine hydrochloride (HCl) and Calcium hydroxylapatite particles suspended in an aqueous-based gel carrier without 3% lidocaine hydrochloride (HCl)
Period: Overall Study
Arm/Group | Radiesse® Mixed With Lidocaine and Radiesse® Without Lidocaine
Started | 102
Completed | 101 (One subject's treatment fold not injected due to adverse event during control fold injection)
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Radiesse® Mixed With Lidocaine and Radiesse® Without Lidocaine
Number analyzed (Participants) | 102
Age, Customized [Mean (Standard Deviation); unit: years] | 48.85 (9.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87
  Male | 15
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 88
  African American | 8
  Hispanic | 2
  Asian | 1
  Other | 3
Region of Enrollment [Number; unit: participants]
  Canada | 102
Fitzpatrick Skin Type [Number; unit: participants] — The Fitzpatrick Skin Types (FST) represent a standard classification of skin color based on one's response to sun exposure (i.e., burns or tans), rather than defined by race or ethnicity.
  All FST were eligible for participation in the current study.
  See full FST descriptions in Astner S, Anderson RR. Skin phototypes 2003. J Invest Dermatol. 2004 Feb;122(2):xxx-xxxi.
  participants
    I: burns easily, never tans | 6
    II: burns easily, tans minimally with difficulty | 19
    III: burns moderately, tans moderately & uniformly | 59
    IV: burns minimally, tans moderately & easily | 8
    V: rarely burns, tans profusely | 5
    VI: never burns, tans profusely | 5

OUTCOME MEASURES:

1. Primary Outcome: Pain Score Using a 10-cm Visual Analog Scale (VAS) for Pain (0 = no Pain, 10 = Very Severe Pain)
Description: Assessment of whether a statistically significant reduction in pain score in the Radiesse® Mixed with Lidocaine nasolabial fold was observed when compared to the Radiesse® without Lidocaine nasolabial fold using a 10-cm visual analog pain scale (0 = no pain, 10 = very severe pain).
  In the study protocol, the assessment of achieving a statistically significant reduction in pain at time zero was selected a priori to be analyzed using a paired t-test to test the null hypothesis that the mean of the differences in VAS scores between the Treatment and Control folds is equal to zero.
Time Frame: Immediately after injection (Time 0)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Nasolabial folds
Groups:
- Radiesse® Mixed With Lidocaine: Injectable Dermal Filler. The same participants received the experimental device and the active comparator device at the same time (left and right sides of face).
  Calcium hydroxylapatite particles suspended in an aqueous-based gel carrier containing 3% lidocaine hydrochloride (HCl)
- Radiesse® Without Lidocaine: Injectable Dermal Filler. The same participants received the experimental device and the active comparator device at the same time (left and right sides of face).
  Calcium hydroxylapatite particles suspended in an aqueous-based gel carrier without 3% lidocaine hydrochloride (HCl)
Arm/Group | Radiesse® Mixed With Lidocaine | Radiesse® Without Lidocaine
Number analyzed (Participants) | 101 | 101
Number analyzed (Nasolabial folds) | 101 | 101
units on a scale | 2.32 (1.57) | 6.73 (2.22)
Statistical Analysis 1: Comparison: Radiesse® Mixed With Lidocaine vs Radiesse® Without Lidocaine; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Paired t-test; Mean Difference (Net) = -4.41

2. Secondary Outcome: Number of Participants With a Clinically Meaningful Reduction in Pain As Defined by a ≥ 2.0-cm Reduction in VAS
Description: In this split-face study, a clinically meaningful difference in pain was defined as a 2-cm "reduction" (i.e., subject reports at least 2-cm less pain on a 10-cm VAS) in the Radiesse® Mixed with Lidocaine NLF when compared to the Radiesse® without Lidocaine NLF.
Time Frame: Immediately after injection (Time 0)
Population: In this split-face study, participants received both treatments (i.e., 1 NLF with Radiesse Mixed with Lidocaine and 1 NLF with Radiesse without Lidocaine). Results are presented as the number of participants reporting at least a 2-cm lower pain VAS score in the Radiesse Mixed with Lidocaine NLF when compared to the Radiesse without Lidocaine NLF.
Measure: Number; unit: participants
Groups:
- Radiesse® Mixed With Lidocaine and Radiesse® Without Lidocaine: Injectable Dermal Filler. The same participants received the experimental device and the active comparator device at the same time (left and right sides of face).
  Calcium hydroxylapatite particles suspended in an aqueous-based gel carrier containing 3% lidocaine hydrochloride (HCl) and calcium hydroxylapatite particles suspended in an aqueous-based gel carrier without 3% lidocaine hydrochloride (HCl)
Arm/Group | Radiesse® Mixed With Lidocaine and Radiesse® Without Lidocaine
Number analyzed (Participants) | 101
participants | 91
Statistical Analysis 1: Comparison: Radiesse® Mixed With Lidocaine and Radiesse® Without Lidocaine; 91 (90.1%) of 101 subjects had a ≥ 2.0 cm lower VAS Score in treatment versus control NLF at Time 0; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Binomial proportion, two-sided Fisher's exact test

3. Secondary Outcome: Visual Analogue Scale (VAS) Pain Score 15 Minutes Post Injection
Description: A 10-cm VAS (with 21 total circles, marked at 0.5 cm intervals) was used in which 0 = no pain and 10 = very severe pain.
Time Frame: 15 minutes post injection
Population: One subject did not receive treatment in the Radiesse® Mixed with Lidocaine (treatment) fold due to adverse event during injection of the Radiesse® without Lidocaine (control) nasolabial fold, which was randomized to be treated first. This subject was followed through the end of the trial for safety, but was excluded from comparative analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Radiesse® Mixed With Lidocaine | Radiesse® Without Lidocaine
Number analyzed (Participants) | 101 | 101
units on a scale | 1.06 (1.23) | 3.45 (2.31)
Statistical Analysis 1: Comparison: Radiesse® Mixed With Lidocaine vs Radiesse® Without Lidocaine; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Paired t-test

4. Secondary Outcome: Visual Analogue Scale (VAS) Pain Score 30 Minutes Post Injection
Description: A 10-cm VAS (with 21 total circles, marked at 0.5 cm intervals) was used in which 0 = no pain and 10 = very severe pain.
Time Frame: 30 minutes post injection
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Radiesse® Mixed With Lidocaine | Radiesse® Without Lidocaine
Number analyzed (Participants) | 101 | 101
units on a scale | 0.73 (0.99) | 2.52 (2.35)
Statistical Analysis 1: Comparison: Radiesse® Mixed With Lidocaine vs Radiesse® Without Lidocaine; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Paired t-test

5. Secondary Outcome: Visual Analogue Scale (VAS) Pain Score 45 Minutes Post Injection
Description: A 10-cm VAS (with 21 total circles, marked at 0.5 cm intervals) was used in which 0 = no pain and 10 = very severe pain.
Time Frame: 45 minutes post injection
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Radiesse® Mixed With Lidocaine | Radiesse® Without Lidocaine
Number analyzed (Participants) | 101 | 101
units on a scale | 0.48 (0.78) | 1.78 (2.00)
Statistical Analysis 1: Comparison: Radiesse® Mixed With Lidocaine vs Radiesse® Without Lidocaine; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Paired t-test

6. Secondary Outcome: Visual Analogue Scale (VAS) Pain Score 60 Minutes Post Injection
Description: A 10-cm VAS (with 21 total circles, marked at 0.5 cm intervals) was used in which 0 = no pain and 10 = very severe pain.
Time Frame: 60 minutes post injection
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Radiesse® Mixed With Lidocaine | Radiesse® Without Lidocaine
Number analyzed (Participants) | 101 | 101
units on a scale | 0.31 (0.66) | 1.09 (1.56)
Statistical Analysis 1: Comparison: Radiesse® Mixed With Lidocaine vs Radiesse® Without Lidocaine; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Paired t-test

7. Secondary Outcome: Visual Analogue Scale (VAS) Pain Score 1 Week Post Injection
Description: A 10-cm VAS (with 21 total circles, marked at 0.5 cm intervals) was used in which 0 = no pain and 10 = very severe pain.
Time Frame: 1 week post injection
Population: Two subjects missed their Week 1 visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Radiesse® Mixed With Lidocaine | Radiesse® Without Lidocaine
Number analyzed (Participants) | 99 | 99
units on a scale | 0.05 (0.32) | 0.04 (0.31)
Statistical Analysis 1: Comparison: Radiesse® Mixed With Lidocaine vs Radiesse® Without Lidocaine; Test type: Superiority or Other; p = 0.5663, t-test, 2 sided — Paired t-test

8. Secondary Outcome: Visual Analogue Scale (VAS) Pain Score 2 Weeks Post Injection
Description: A 10-cm VAS (with 21 total circles, marked at 0.5 cm intervals) was used in which 0 = no pain and 10 = very severe pain.
Time Frame: 2 weeks post injection
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Radiesse® Mixed With Lidocaine | Radiesse® Without Lidocaine
Number analyzed (Participants) | 101 | 101
units on a scale | 0.01 (0) | 0 (0)
Statistical Analysis 1: Comparison: Radiesse® Mixed With Lidocaine vs Radiesse® Without Lidocaine; Test type: Superiority or Other; p = 0.3197, t-test, 2 sided — Paired t-test

9. Secondary Outcome: Visual Analogue Scale (VAS) Pain Score 4 Weeks Post Injection
Description: A 10-cm VAS (with 21 total circles, marked at 0.5 cm intervals) was used in which 0 = no pain and 10 = very severe pain.
Time Frame: 4 weeks post injection
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Radiesse® Mixed With Lidocaine | Radiesse® Without Lidocaine
Number analyzed (Participants) | 101 | 101
units on a scale | 0 (0) | 0 (0)

10. Secondary Outcome: Assess Subject Preference to Pain
Description: 2 questions were asked of 101 subjects: 1) Was one treatment less painful than the other? and 2) Was the difference in pain levels significant enough to affect your preference for one treatment over the other?
  Only those participants responding "yes" to these 2 questions about pain and preference for treatment are reported in the table below.
Time Frame: Immediately after injection (Time 0)
Measure: Number; unit: participants responding "yes"
Groups:
- Radiesse® Mixed With Lidocaine and Radiesse® Without Lidocaine: Injectable Dermal Filler. The same participants received the experimental device and the active comparator device at the same time (left and right sides of face).
  Calcium hydroxylapatite particles suspended in an aqueous-based gel carrier containing 3% lidocaine hydrochloride (HCl) and without 3% lidocaine hydrochloride (HCl)
Arm/Group | Radiesse® Mixed With Lidocaine and Radiesse® Without Lidocaine
Number analyzed (Participants) | 101
participants responding "yes"
  Was One Treatment Less Painful Than the Other? | 98
  Pain Significant Enough to Affect Preference? | 87

ADVERSE EVENTS:
Arm/Group | Radiesse® Mixed With Lidocaine | Radiesse® Without Lidocaine
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/101
Other Adverse Events (participants affected / at risk) | 90/101 | 92/101
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiesse® Mixed With Lidocaine (N=101) | Radiesse® Without Lidocaine (N=101)
Bruising (Skin and subcutaneous tissue disorders) | 44 (44) | 48 (48)
Itching (Skin and subcutaneous tissue disorders) | 37 (37) | 34 (34)
Pain (Skin and subcutaneous tissue disorders) | 48 (48) | 57 (57)
Redness (Skin and subcutaneous tissue disorders) | 66 (66) | 71 (71)
Swelling (Skin and subcutaneous tissue disorders) | 90 (90) | 92 (92)
Blanching (Skin and subcutaneous tissue disorders) | 5 (5) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No